CLINICAL TRIAL: NCT04974879
Title: Osimertinib Combined With Bevacizumab in the Treatment Epidermal Growth Factor Receptor (EGFR) Exon 20 Insertions Local Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Osimertinib Combined With Bevacizumab in the Treatment Epidermal Growth Factor Receptor (EGFR) Exon 20 Insertions Metastatic Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Principal Investigator, Youxin Ji, chief, Qingdao Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QDCH2021-07-02
Record Dates: First submitted 2021-07-16; First posted 2021-07-23 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Bronchial Neoplasms; EGFR Exon20ins Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Bronchial Neoplasms | interventions — osimertinib; Bevacizumab

STUDY DESIGN:
Intervention Model Description: osimertinib oral and bevazizumab intravenously
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study drug (Experimental): osimertinib oral daily and bevacizumab 15mg/KG body weight intravenously infusion every 21 days.
  Interventions: Drug: Osimertinib Oral Tablet

INTERVENTIONS:
Drug: Osimertinib Oral Tablet — Osimertinib, 80mg, oral daily; bevacizumab (avastin), 15mg/KG body weight, erery 21 days, intravenously.
  Other Names: bevacizumab

SUMMARY:
There is no muture method to treat EGFR 20 insertion mutation non-small-cell lung cancer (NSCLC). the he purpose of this study is to study osimertinib combined with bevacizumab in the management of it.

DETAILED DESCRIPTION:
Lung cancer is one of the most common types of cancer and is the most common cause of death from cancer (almost 20 percent [%] of cancer deaths); NSCLC accounts for 80% to 85% of lung cancers. The hypothesis is that osimertinib combined bevacizumab in patients with locally advanced or metastatic NSCLC characterized by EGFR Exon 20ins activating mutations. Efficacy assessments will include disease assessment, symptomatic progression and patient-reported outcome. Safety assessments will include physical examinations, vital signs, electrocardiograms (ECGs), Eastern Cooperative Oncology Group (ECOG) performance status and clinical safety laboratory assessments (serum chemistry, hematology, coagulation, and urinalysis).

ELIGIBILITY:
Inclusion Criteria:

Participant must have histologically or cytologically confirmed, locally advanced or metastatic, nonsquamous non-small cell lung cancer (NSCLC) with documented primary epidermal growth factor receptor (EGFR) Exon 20ins activating mutation Participant must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

Participant must have Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1, or 2 Participant must agree to genetic characterization of tumor status through the required pretreatment tumor biopsy (or submission of equivalent archival material), as well as baseline and periodic blood samples for analysis of tumor mutations in the bloodstream A female participant of childbearing potential must have a negative serum or urine test at screening and within 72 hours of the first dose of study treatment and must agree to further serum or urine pregnancy tests during the study

Exclusion Criteria:

Participant has history of spinal cord compression that has not been treated definitively with surgery or radiation Participant has a medical history of interstitial lung disease (ILD), including drug-induced ILD, or radiation pneumonitis Participant has a contraindication to the use Osimertinib or Bevacizumab

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 18 months
  Progression-Free Survival (PFS) According to RECIST v1.1 as Assessed by Blinded Independent Central Review (BICR)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 48 months
  ORR is defined as the percentage of participants who achieve either a complete response (CR) or partial response (PR) as defined by BICR using RECIST v1.1 criteria.
Overall Survival (OS) | Up to 48 months
  Overall Survival is defined as the time from the date of randomization to the date of participant's death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao Central Hospital, Qingdao Cancer Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No